CLINICAL TRIAL: NCT02745587
Title: The N+-PROPER Trial: Evaluating the Impact of Prostate Only Versus Pelvic Radiation for N+ Prostate Cancer.
Brief Title: Evaluating the Impact of Prostate Only Versus Pelvic Radiation for N+ Prostate Cancer.
Acronym: PROPER
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Stopped because of poor accrual in June 2021 after the inclusion of 69 patients
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016/0246
Record Dates: First submitted 2016-04-15; First posted 2016-04-20 (Estimated); Last update posted 2022-12-28 (Actual); Status verified 2016-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prostate(bed) only (Experimental): external beam radiotherapy limited to the prostate(bed)
  Interventions: Radiation: radiotherapy
- Prostate(bed) and pelvis (Active Comparator): external beam radiotherapy to the prostate(bed) and pelvic lymph node regions
  Interventions: Radiation: radiotherapy

INTERVENTIONS:
Radiation: radiotherapy — high dose external beam radiotherapy limited to the prostate(bed)

SUMMARY:
At least 40% of the patients with prostate cancer (PC) present with positive lymph nodes (N1). The optimal treatment strategy for these patients remains controversial. Although androgen deprivation therapy (ADT) is still often initiated as only treatment, the results are disappointing. Recent studies support the use of more aggressive therapies including external beam radiotherapy (EBRT) and ADT. The retrospective studies supporting the additional use of EBRT in N1 PC patients are however not conclusive regarding to the extent of radiation field.

Even after an EPLND, there might be a role for pelvic EBRT in irradicating microscopic disease. However pelvic irradiation irrevocably results in increased toxicity. Moreover, in node negative (N0) PC patients the addition of pelvic EBRT has not resulted in improved outcome in randomised trials. However in the setting of Tumor Node Metastasis pathological stage (p)N1, proven on pathological examination, PC patients this has never been evaluated so far. This trial aims to answer the question whether or not pelvic EBRT is beneficial in pathological N1 PC patients. It is also important to realise that not all pathological N1 PC patients have similar outcome. There is a significant impact of number of positive lymph nodes on outcome, with two positive nodes being suggested as a significant cut-off value in predicting survival in pathological N1 PC patients. By stratifying the patients according to the number of lymph nodes involved this study will add to the proper selection of those patients who will benefit most of pelvic EBRT and avoid toxicity in patients who have no benefit of pelvic EBRT.

Additionally, small RNAs constitute potentially valuable markers for the diagnosis, prognosis, and therapeutic choices in PC patients. Blood samples will be collected to examine the potential role of miRNAs as a biomarker and to develop a prognostic signature for clinical relapse-free survival.

The results of this trial will serve as a base for developping new trials in order to optimise the treatment of patients with pathological N1 PC.

DETAILED DESCRIPTION:
In an era with increasing evidence in favour of an aggressive local treatment, where an extended pelvic lymph node dissection (EPLND) is more frequently performed and with data supporting the potential role for external beam radiotherapy (EBRT) in pelvic node positive (N1) prostate cancer (PC), the treatment of N1 PC patients needs to be revised. Seen the lack of clear guidelines regarding the extent of radiation field in N1 prostate cancer patients, there is an urgent need for studies evaluating the place of pelvic EBRT.

The aim of this trial is thus to evaluate if pelvic irradiation has an impact on clinical relapse free survival in pathological N1 PC.

The hypothesis is that performing a pelvic EBRT after EPLND in pathological N1 PC patients results in a significant improved clinical relapse free survival with 15% when compared to prostate only EBRT.

This will be evaluated in a multicentre Phase III stratified randomised trial randomising patients with PC and 1-4 positive lymph nodes on EPLND between prostate(bed) only radiotherapy + 2 years of ADT or pelvic radiotherapy + 2 years of androgen deprivation. A total of 330 patients will be enrolled in this trial. Stratification is based on the number of positive lymph nodes since patients with increased number of positive lymph nodes exhibit a poorer prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Histological proven carcinoma of the prostate
* Positive lymph nodes found on extended pelvic dissection (EPLND) defined as:
* Removal of the lymphatic tissue in the obturator fossa + along the external iliac vessels + additional complete resection of the lymph nodes (lnn) along, medially and laterally to, the hypogastric vessels
* If technically feasible: removal of lnn along the common iliac vessels
* Removal of ≥10 lnn
* Treatment of the primary tumor by either radical prostatectomy or EBRT
* Willing to receive androgen deprivation therapy
* World health organization 0-2
* Written informed consent

Exclusion Criteria:• >4 positive lnn found on EPLND

* Prior pelvic irradiation
* Other primary tumor (except for non-melanoma skin tumors) diagnosed <5 years before enrollment
* Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2022-09-22 (Actual)

PRIMARY OUTCOMES:
Assessment of number of participants without clinical relapse | 8 years
  presence of loco(regional) release or distant metastases

SECONDARY OUTCOMES:
Assessment of number of participants experiencing Radiation Therapy Oncology Group toxicity | 5 years
  acute
Assessment of number of participants experiencing Radiation Therapy Oncology Group toxicity | 10 years
  late
Assessment of number of participants with biochemical control | 8 years
  absence of prostate specific antigen relapse

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Fonteyne, Prof, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided